CLINICAL TRIAL: NCT00883662
Title: Mirena Observational Program
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14474; MA0910KZ (Other: company internal)
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Contraception; Menorrhagia; Endometrial Hyperplasia; Estrogen Replacement Therapy
MeSH Terms: conditions — Menorrhagia; Endometrial Hyperplasia | interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Levonorgestrel (Mirena, BAY86-5028)

INTERVENTIONS:
Drug: Levonorgestrel (Mirena, BAY86-5028) — Patients older than 18 years with previously taken decision of their gynecologist to insert Mirena according to registered indications

SUMMARY:
Mirena is used for long-term in Kazakhstan, and in our observational program we would like to study patients distribution per indications of Mirena, and also patient compliance within a year after Mirena insertion. For patients with all approved indications for Mirena use: contraception, treatment of menorrhagia and protection from endometrial hyperplasia during estrogen replacement therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with previously taken decision of their gynecologist to insert Mirena according to registered indications

Exclusion Criteria:

* All patients with contraindications to Mirena insertion, according to approved prescribing information.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years with previously taken decision of their gynecologist to insert Mirena according to registered indications
Sampling Method: Non-Probability Sample
Enrollment: 2725 (Actual)
Dates: Start 2009-05; Primary Completion 2014-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Patient distribution per indication | 12 months

SECONDARY OUTCOMES:
Patient compliance | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Kazakhstan